CLINICAL TRIAL: NCT06006013
Title: Phase II Open Label, Single-Arm Study of Cabozantinib in Combination With Pembrolizumab in the Treatment of Locally Advanced or Metastatic Adrenocortical Carcinoma
Brief Title: Cabozantinib in Combination With Pembrolizumab for the Treatment of Patients With Locally Advanced, Metastatic, or Unresectable Adrenal Cortical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bassel Nazha, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005532; NCI-2023-04952 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00005532 (Other: Emory University); WINSHIP5823-22 (Other: Emory University); P30CA138292 (NIH)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Adrenal Cortex Carcinoma; Adrenal Cortical Carcinoma; Stage III Adrenal Cortex Carcinoma; Stage IV Adrenal Cortex Carcinoma AJCC v8; Unresectable Adrenal Cortex Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Cortex Neoplasms | interventions — pembrolizumab; Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cabozantinib, pembrolizumab) (Experimental): Patients receive cabozantinib orally (PO) once daily (QD) on days 1-21 of each cycle and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) at screening and then every 12 weeks on study and undergo collection of blood samples at screening, on study, and at end of treatment. Patients without archival tissue also undergo biopsy at screening.
  Interventions: Biological: Pembrolizumab; Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: KEYTRUDA
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: Cabometyx; Cometriq
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase II trial tests how well cabozantinib in combination with pembrolizumab works in treating patients with adrenocortical cancer that has spread to nearby tissue or lymph nodes (locally advanced), that has spread from where it first started (primary site) to other places in the body (metastatic), or that cannot be removed by surgery (unresectable). Cabozantinib inhibits receptor tyrosine kinases, which are receptors commonly over-expressed by tumor cells. This may result in an inhibition of both tumor growth and blood vessel formation, eventually leading to a decrease in tumor size or extent in the body. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Adding cabozantinib to pembrolizumab may be more effective at treating patients with adrenal cortical cancer than giving these drugs alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the anti-tumor activity of the combination of cabozantinib S-malate (cabozantinib) and pembrolizumab by assessing the overall response rate (ORR) as measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1.).

SECONDARY OBJECTIVE:

I. To evaluate the efficacy of the combination of cabozantinib and pembrolizumab as measured by progression free survival and overall survival assessed up to 2 years, safety and tolerability of the combination.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To assess tissue-based assays in archival tissue and correlative changes in peripheral T-cell subsets, myeloid derived suppressor cells (MDSC), blood inflammatory markers and cytokines.

OUTLINE:

Patients receive cabozantinib orally (PO) once daily (QD) on days 1-21 of each cycle and Pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) at screening and then every 12 weeks on study and undergo collection of blood samples at screening, on study, and at end of treatment. Patients without archival tissue also undergo biopsy at screening.

After completion of study treatment, patients are followed for 28 days and then up to 2 years

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 ,Karnofsky >= 50%.
* Metastatic disease or unresectable locally advanced disease.
* Histologically documented adrenal cortical carcinoma.
* Untreated or having received any number of lines of prior therapy.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Life expectancy >= 12 weeks
* Tumor tissue samples must be available for submission prior to initiation of study treatment. If not, agree to undergo biopsy.
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version 5 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically nonsignificant and/or stable on supportive therapy.
* Absolute neutrophil count (ANC) >= 1500/uL without granulocyte colony-stimulating factor support within 28 days before first dose of study treatment.
* Lymphocyte count 0.5 x 10^9/L (500/mL) within 28 days before first dose of study treatment.
* White blood cell count >= 2500/uL within 28 days before first dose of study treatment.
* Platelets >= 100,000/uL without transfusion within 28 days before first dose of study treatment.
* Hemoglobin >= 9 g/dL (>= 90 g/L). Patients may be transfused to meet this criterion within 28 days before first dose of study treatment.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) =< 3 x upper limit of normal (ULN). ALP =< 5 x ULN with documented bone metastases within 28 days before first dose of study treatment.
* Total bilirubin =< 1.5 x ULN for subjects with Gilbert's disease =< 3 x ULN within 28 days before first dose of study treatment.
* Serum albumin >= 2.8 g/dl within 28 days before first dose of study treatment.
* Prothrombin time (PT) / international normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN within 28 days before first dose of study treatment.
* Serum creatinine =< 1.5 x ULN or calculated creatinine clearance >= 40mL/min (>= 0.675mL/sec) using the Cockcroft-Gault equation within 28 days before first dose of study treatment.
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg (=< 113.2 mg/mmol), or 24-h urine protein =< 1 g within 28 days before first dose of study treatment.
* Negative human immunodeficiency virus (HIV) test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/uL, and have an undetectable viral load.
* Negative hepatitis B surface antigen (HBsAg) test at screening.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative hepatitis C virus (HCV) ribonucleic acid (RNA) test at screening.

  * The hepatitis C virus (HCV) ribonucleic acid (RNA) test must be performed for patients who have a positive HCV antibody test
* The effects of study drugs on the developing human fetus are unknown. For this reason, female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* Female of child-bearing potential (FCBP) and men treated or enrolled on this protocol must agree to use adequate contraception with a failure rate < 1% prior to study entry, for the duration of study participation, and 5 months after completion of study drug administration.

  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence e.g., calendar, ovulation, symptothermal, or postovulation methods and withdrawal are not adequate methods of contraception
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating [FSH] level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Receipt of any type of small molecule kinase inhibitor including investigational kinase inhibitor within 2 weeks before first dose of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including immunostimulatory agents or investigational agents) within 4 weeks or 5 half-lives of the drug (whichever is longer) before first dose of study treatment
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects with known brain metastases or cranial epidural disease should also have no history of intracranial hemorrhage or spinal hemorrhage. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment. If subject is receiving anti-convulsant therapy, the dose is considered stable
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH)
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Administration of a live, attenuated vaccine within 30 days before first dose of study treatment or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Concomitant mitotane use

  * Mitotane must have been discontinued 28 days prior to first dose of study treatment, with mitotane serum level < 2 mg/L if mitotane administered within last 6 months
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment
    * Stroke, including transient ischemic attack (TIA), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment

      * Subjects with a diagnosis of incidental, subsegmental pulmonary embolism (PE) or deep vein thrombosis (DVT) within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
  * Uncontrolled tumor-related pain:

    * Patients requiring pain medication must be on a stable regimen at study entry
    * Symptomatic lesions e.g., bone metastases or metastases causing nerve impingement amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation (see exclusion criteria #4 for minimal required duration prior to trial enrollment)
    * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
  * Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

    * Patients with indwelling catheters (e.g., PleurX) are allowed
  * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

    * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Lesions invading or encasing any major blood vessels
* Other clinically significant disorders that would preclude safe study participation.

  * Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

    * Type 1 diabetes mellitus on an insulin regimen
    * Hypothyroidism only requiring hormone replacement
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF]-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after principal investigator confirmation has been obtained
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma or mitotane-associated adrenal insufficiency, or low-dose corticosteroids for orthostatic hypotension or other causes of adrenal insufficiency are eligible for the study
    * Inhaled, intranasal, intra-articular, or topical steroids are permitted
  * Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
  * Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
  * History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

    * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
  * Serious non-healing wound/ulcer/bone fracture
  * Malabsorption syndrome
  * Uncompensated/symptomatic hypothyroidism
  * Moderate to severe hepatic impairment (Child-Pugh B or C)
  * Requirement for hemodialysis or peritoneal dialysis
  * History of solid organ or allogenic stem cell transplant
  * Known history of COVID-19 unless the subject has clinically recovered from the disease at least 30 days prior to first dose of study treatment
  * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. Furthermore, subjects with a history of additional risk factors for torsades de pointes (e.g., long QT syndrome) are also excluded. Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Pregnant or lactating females
* Inability to swallow tablets or unwillingness or inability to receive IV administration
* Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Current treatment with anti-viral therapy for hepatitis B virus (HBV).
* History of leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Every 12 weeks, assessed up to 2 years
  Overall response rate is defined as the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors version 1.1. Overall response rate will be estimated by the Clopper-Pearson method with 95% confidence intervals. Descriptive statistics on continuous data will include means, medians, standard deviations, and ranges, while categorical data will be summarized using frequency counts and percentages. Will explore whether the sample size can inform on the association between overall response rate and demographics or molecular biomarkers by Fisher's exact test -categorical variables and Wilcoxon rank-sum test -continuous variables, wherever appropriate this analysis is exploratory in nature.

SECONDARY OUTCOMES:
Progression free survival | From treatment initiation until disease progression, death due to disease, or lost to follow up, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate median event time with 95% confidence interval.
Overall survival | From treatment initiation until death due to any cause or loss to follow up, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate median event time with 95% confidence interval.
Incidence of adverse events | Up to 2 years
  Evaluated according to the Common Terminology Criteria for Adverse Events version 5.0. Safety endpoints will be tabulated using frequency such as percent with at least one adverse event, percent for each grade, and percent with grade 3 or more adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bassel Nazha, MD, MPH, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia